CLINICAL TRIAL: NCT02883296
Title: Long-term Follow-up of Anal Fistulae in Crohn's Disease Treated With Anti-TNFalpha and Interest of New MRI Sequences
Acronym: FISTULE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2010-A00588-31
Record Dates: First submitted 2016-08-23; First posted 2016-08-30 (Estimated); Last update posted 2021-04-28 (Actual); Status verified 2016-08

CONDITIONS: Anal Fistula; Crohn's Disease
MeSH Terms: conditions — Rectal Fistula; Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients with perianal fistulizing Crohn's disease (Experimental)
  Interventions: Other: Pelvis Magnetic resonance imaging

INTERVENTIONS:
Other: Pelvis Magnetic resonance imaging

SUMMARY:
Main purposes of this study are :

* Analysis of relapse risk of anal fistulae with prospective follow-up of patients undergoing pelvic MRI every 6 months for one year. This monitoring also determines if the presence of path of fistulae visible on MRI during inclusion visit is associated to increased risk of perianal abscess under infliximab or adalimumab treatment.
* Evaluation of interest of new magnetic resonance imaging sequences for detection of persistent anal fistulae under infliximab or adalimumab treatment.

Secondary purposes are:

* Description of patients with one or more paths of fistulae visible with MRI after at least one year of treatment with infliximab or adalimumab administered for anal fistulae and showing a complete healing of fistulae at clinical examination of inclusion visit.
* Identification of predictive factors (included the presence of paths of fistulae visible with MRI during inclusion visit) of relapse of anal fistulae during the 1-year-follow-up after inclusion visit.

ELIGIBILITY:
Inclusion Criteria:

* Aware and cooperative, giving written consent
* Crohn's disease diagnosed with clinical, biological, endoscopic and/or radiologic criteria
* Patient treated with infliximab or adalimumab for perianal fistulizing Crohn's disease since at least one year
* Absence of drainage seton at inclusion
* Absence of active perianal lesions at inclusion: absence of suggestive symptoms and normal proctologic clinical examination without general anesthesia
* Patient with MRI monitoring for perianal fistulizing Crohn's disease

Exclusion Criteria:

* Patient under juridical protection or without affiliation to social security
* Refusal or impossibility of giving informed consent
* Patient not followed-up by MRI or having a contraindication for MRI, especially the presence of cardiac stimulators or implantable defibrillators, cochlear implants, neurosurgical clips, intra-orbital or encephalic metallic foreign bodies, endo-prostheses placed since at least 4 weeks or osteosynthesis material placed since less than 6 weeks or gadolinium intolerance history
* Surgery for Crohn's disease already planned at inclusion visit, individual participating to another study evaluating efficacy and/or tolerance of medical or surgical treatment for perianal fistulae of Crohn's disease
* Patient treated with anti-TNF for luminal Crohn's disease
* Patient having active perineal lesions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Evaluation of severity of Crohn's disease with Van Assche MRI score | day 0
Evaluation of severity of Crohn's disease with Van Assche MRI score | 6 months
Evaluation of severity of Crohn's disease with Van Assche MRI score | 1 year

SECONDARY OUTCOMES:
Evaluation of activity of Crohn's disease with CDAI score | day 0
Evaluation of activity of Crohn's disease with CDAI score | 6 months
Evaluation of activity of Crohn's disease with CDAI score | 1 year
Evaluation of severity of perianal injury with PDAI score | day 0
Evaluation of severity of perianal injury with PDAI score | 6 months
Evaluation of severity of perianal injury with PDAI score | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Peyrin-Biroulet, Pr, Principal Investigator — Service d'Hépato Gastro-entérologie Hôpital BRABOIS- CHU de NANCY

IPD SHARING:
Plan to Share IPD: No